CLINICAL TRIAL: NCT06724549
Title: A Study to Evaluate the Effect of Food on the Pharmacokinetics of BN104 Tablets in Healthy Subjects
Brief Title: The Effect of Food on the Pharmacokinetics of BN104 Tablets
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: BioNova Pharmaceuticals (Shanghai) LTD. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: BN104-106
Record Dates: First submitted 2024-12-02; First posted 2024-12-09 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2024-12

CONDITIONS: Health Subjects

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Fasting-Fed (Active Comparator): Patients will be administrated 600mg dose of BN104 tablets under fasting conditions and fed conditions in period 1 and 2 respectively. There will be a at least 7-day washout period between the first and second dose.
  Interventions: Drug: BN104
- Fed-Fasting (Active Comparator): Patients will be administrated 600mg dose of BN104 tablets under fed conditions and fasting conditions in period 1 and 2 respectively. There will be a at least 7-day washout period between the first and second dose.
  Interventions: Drug: BN104

INTERVENTIONS:
Drug: BN104 — This study adopts two-treatment (fasting or following a high-fat meal), two-period, two-sequence crossover design. The subjects will be randomly assigned into one of two treatment sequences in a 1:1 ratio. A single 600 mg dose of BN104 tablets administered under fasting conditions or after a standard high-fat breakfast in period 1 and 2.

SUMMARY:
The goal of the clinical trial is to evaluate the effect of food on the Pharmacokinetics of BN104 tablets in healthy subjects. The main questions it aims to answer are:

Whether the pharmacokinetic characteristics of BN104 tablets will be affected by food? How well is the safety and tolerability of BN104 tablets in healthy subjects? To preliminarily evaluate the effect of BN104 on the QTc interval.

DETAILED DESCRIPTION:
This study adopted a single-center, randomized, open-label, single-dose, two-treatment (fasting or following a high-fat meal), two-period, and two-sequence crossover design. A total of 16 healthy subjects were enrolled in this trial. The subjects were randomized two days before dosing, and the subjects were randomly assigned to the fasting to high-fat meal group or the high-fat meal to fasting group with 8 subjects in each group. The single-dose regimen was adopted in this study, and the washout period between the periods was 7 days.

ELIGIBILITY:
Inclusion:

1. Age ≥ 18 years, male or female;
2. Male subjects weighed ≥ 50.0 kg and female subjects weighed ≥45.0 kg, with a body mass index (BMI) between 19 and 26 kg/m2 (both inclusive);
3. Subjects must fully understand the purpose, nature, methods, and potential adverse reactions of the study and voluntarily consent to participate. Prior to any study procedures, subjects must provide written informed consent and ensure their personal participation in all study-related procedures.

Exclusion Criteria:

1. (Inquiry) A history or current presence of clinically significant diseases affecting the circulatory, endocrine, nervous, gastrointestinal, respiratory systems, or hematologic, immunologic, psychiatric, or metabolic disorders, or any other conditions (e.g., heart failure, hypokalemia, hypomagnesemia, family history of long QT syndrome) that could interfere with study outcomes;
2. (Inquiry) Those who have any history of allergy to two or more drugs, food, or other substances, or are allergic to any of the components of the investigational drug;
3. (Inquiry) Those who have undergone surgery within 28 days prior to the first dose of the investigational drug or who plan to have surgery during the trial;
4. (Inquiry) Those who have been vaccinated 1 month before the first administration of the investigational drug, or those who plan to be vaccinated during the trial;
5. (Inquiry) Those who have received any medications or health care products (including Chinese Herbal Medicine) within 14 days prior to the first dose of the investigational drug;
6. (Inquiry) Use of any drugs that may influence the pharmacokinetics of the investigational drug within 30 days prior to the first dose, including: strong CYP3A4 inhibitors: e.g., ketoconazole, itraconazole, clarithromycin, atazanavir, ritonavir, indinavir, voriconazole; moderate CYP3A4 and/or P-glycoprotein (P-gp) inhibitors: e.g., fosamprenavir, aprepitant, erythromycin, fluconazole, verapamil, diltiazem; strong CYP3A4 inducers: e.g., phenytoin, carbamazepine, rifampin, rifabutin, rifapentine, phenobarbital, and St. John's wort;
7. (Inquiry) Those who have received any clinical trial drug or enrolled in any drug/medical device clinical trial within 3 months prior to the first dose of investigational drug;
8. (Inquiry) Blood donors who have donated blood within 3 months prior to the first dose of investigational drug, or those who have lost more than 400 mL of blood within 3 months prior to the first dose of investigational drug;
9. (Inquiry) Individuals who cannot tolerate venipuncture and/or have a history of blood and needle sickness;
10. (Inquiry) Those who have received oral contraceptives within 30 days prior to the first dose of investigational drug or who have received long-acting estrogen or progestin injections or implants within 6 months prior to the first dose of investigational drug;
11. (Inquiry) Those who have had unprotected sex within 14 days prior to the first dose of the investigational drug (females), or females who are pregnant or breastfeeding;
12. (Inquiry) Those who cannot take at least 1 non-medication contraceptive measure with the partner throughout the trial, or those who plan to bear a child, donate sperm, or donate egg within 3 months after the study completion;
13. (Inquiry) Those who have special requirements for diet and cannot follow a unified diet;
14. (Inquiry) Those with dysphagia;
15. (Inquiry) Those who have consumed excessive amounts of tea, coffee, or caffeinated beverages (more than 8 cups, 1 cup = 250 mL) per day during the 3 months prior to the first dose of the investigational drug;
16. (Inquiry) Those who have ingested or plan to ingest any caffeine-containing foods or beverages (e.g., coffee, strong tea, chocolate, etc.) or foods (e.g., sardines, animal livers, etc.) or beverages that are rich in xanthine components within 48 hours prior to the first dose of study drug;
17. (Inquiry) Those who have consumed foods that can affect the in vivo metabolism of the drug (including citrus fruits such as grapefruit, lime, and pomelo, and pitaya, mango, carambola, papaya, and pomegranate, etc.), or other foods that can affect drug absorption, distribution, metabolism, or excretion within 7 days before the first dose of the investigational drug and considered as not suitable to participate in the trial by the investigator; or those who refuse to discontinue such diet during the trial;
18. (Inquiry) Addicted to smoking, daily smoking of more than five cigarettes within three months prior to the first dose, or inability to discontinue smoking of any tobacco products during this trial;
19. (Inquiry) Alcoholics or regular drinkers within the 6 months before the first dose of the investigational drug, i.e., more than 14 units of alcohol per week (1 unit of ≈ 200 mL of beer with 5% alcohol content or 25 mL of spirits with 40% alcohol content or 85 mL of wine with 12% alcohol content), or those unable to abstain from alcohol during the study;
20. Screening results showing ALT > 1.5×ULN and/or AST > 1.5×ULN and/or bilirubin > 1.5×ULN for liver function and/or creatinine > 1.0×ULN for renal function;
21. ECG results at screening showing QTcF > 450 ms (calculated using Fridericia's formula: QTcF = QT/(RR)1/3);
22. Those with any clinically significant abnormalities in vital signs, physical examination, ECG, or laboratory tests, as judged by the study doctor, that could pose increased safety risks if participating in the study.
23. Those who may not be able to complete this trial for other reasons or who shall not be included in the opinion of the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2025-01-12 (Actual); Primary Completion 2025-02-13 (Actual); Study Completion 2025-02-13 (Actual)

PRIMARY OUTCOMES:
Peak concentration (Cmax) | 2 weeks
  Assess the Cmax of BN104 and its metabolite BNM-1263
Auc(0-last） | 2 weeks
  Assess the area under the plasma concentration-time curve from time zero to the last quantifiable time point of BN104 and its metabolite BNM-1263
Auc(0-∞） | 2 weeks
  Assess the area under the plasma concentration-time curve from time zero to infinity of BN104 and its metabolite BNM-1263

SECONDARY OUTCOMES:
Time to maximum concentration (Tmax) | 2 weeks
  Assess the Tmax parameters of BN104 and its metabolite BNM-1263
Elimination half-life (t½) | 2 weeks
  Assess the elimination half-life (t½) parameters of BN104 and its metabolite BNM-1263
apparent clearance (CL/F) | 2 weeks
  Assess the apparent clearance (CL/F) parameters of BN104 and its metabolite BNM-1263
apparent volume of distribution (Vz/F) | 2 weeks
  Assess the apparent volume of distribution (Vz/F) parameters of BN104 and its metabolite BNM-1263
adverse events (AEs) | 2 months
  Assess the incidence and grade of AEs
12-lead electrocardiograms (ECGs) | 2 months
  Assess the correlation between plasma concentrations of BN104 and QTc interval.

CONTACTS AND LOCATIONS:
Locations (1):
- Xiangya Hospital of Central South University, Changsha, Hunan, China